CLINICAL TRIAL: NCT03518931
Title: Understanding Fitness' Function in Determining Activity
Acronym: UFFDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1406M51128
Record Dates: First submitted 2018-04-05; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Exercise; Fitness; Strength
MeSH Terms: conditions — Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This arm included individuals randomized to receiving fitness information only.
- Intervention (Experimental): This arm included individuals randomized to having fitness assessments performed.
  Interventions: Diagnostic Test: Fitness testing

INTERVENTIONS:
Diagnostic Test: Fitness testing — The intervention in this study was measuring cardiorespiratory fitness and muscular strength and providing normative data to subjects.
  Arms: Intervention

SUMMARY:
The purpose of the study is to determine how measuring strength (by squeezing a tool called a hand grip dynamometer) and cardiorespiratory fitness (by climbing stairs) and sharing the results with subjects impacts exercise.

DETAILED DESCRIPTION:
The Understanding Fitness Function in Determining Activity (UFFDA) Study was initiated at the 2014 and 2015 Minnesota State Fair to determine if measuring muscular strength and CRF would motivate individuals to increase their physical activity. Eligible individuals consented to participate and were randomized in a 1:1 allocation to control or intervention groups. All participants provided their current Exercise Vital Sign (EVS calculated by multiplying the number of moderate-vigorous exercise sessions/week by the average minutes/session). The intervention group had VO2max estimated using a timed previously validated Step Test and muscular strength measured using a Hand Dynamometer. Results with age appropriate normative data for both grip strength and a "good or superior" VO2max were provided to the intervention group. Our hypothesis was participants who receive the intervention would increase physical activity (measured by EVS) compared to control participants.

ELIGIBILITY:
Inclusion Criteria:

Greater then 18 years old and able to complete the 20-step test to estimate CRF.

Exclusion Criteria:

History of heart disease, Syncope, Chest pain, Dyspnea, Use of beta blockers, Use of non-dihydropyridine calcium channel blockers, Evidence of any unstable medical conditions. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1315 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Exercise vital sign | Baseline to 1 year
  The primary outcome of the study was change in exercise vital sign: (EVS calculated by multiplying the number of moderate-vigorous exercise sessions/week by the average minutes/session)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Olson, MD, Principal Investigator — University of Minnesta

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Langland JT, Sathnur N, Wang Q, Olson APJ. Do assessments of cardiorespiratory and muscular fitness influence subsequent reported physical activity? A randomized controlled trial. BMC Sports Sci Med Rehabil. 2021 Jun 15;13(1):69. doi: 10.1186/s13102-021-00295-z. PMID 34130756